CLINICAL TRIAL: NCT06547359
Title: A Study to Evaluate Drug-Drug Interactions of Obicetrapib Tablets and Ezetimibe Tablets in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NewAmsterdam Pharma (Industry)
Collaborators: Pharma Medica Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TA-8995-14
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Ezetimibe

STUDY DESIGN:
Intervention Model Description: Open-label, two-cohort, fixed-sequence, drug-drug interaction study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- obicetrapib with and without co-administration of ezetimibe (Active Comparator): Ezetimibe 10mg tablets daily from Days 1-17 plus obicetrapib 10mg tablets on Day -9 and Day 8
  Interventions: Drug: Obicetrapib 10mg; Drug: Ezetimibe 10mg
- ezetimibe with and without co-administration of obicetrapib (Active Comparator): Obicetrapib 10mg tablets daily from Days 1-15 plus ezetimibe10mg tablets on Day -3 and Day 12
  Interventions: Drug: Obicetrapib 10mg; Drug: Ezetimibe 10mg

INTERVENTIONS:
Drug: Obicetrapib 10mg — tablets
Drug: Ezetimibe 10mg — tablets

SUMMARY:
A Study to Evaluate Drug-Drug Interactions of Obicetrapib Tablets and Ezetimibe Tablets in Healthy Adult Subjects

DETAILED DESCRIPTION:
A Study to Evaluate the PK of obicetrapib tablets with and without co-administration of daily doses of ezetimibe tablets and the PK of ezetimibe tablets with and without co-administration of daily doses of obicetrapib tablets.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking, male and female subjects, from 18 to 65 years of age.
* BMI ≥18.5 and ≥30 kg/m2
* Females may be of childbearing or non-childbearing potential. Childbearing potential (physically capable of becoming pregnant). Non-childbearing potential: Surgically sterile (i.e., both ovaries removed, uterus removed, or bilateral tubal ligation); and/or postmenopausal (no menstrual period for at least 12 consecutive months without any other medical cause and FSH and LH values consistent with being postmenopausal).
* Willing to use acceptable, effective methods of contraception.
* Able to tolerate venipuncture.
* Be informed of the nature of the study and give written consent prior to any study procedure.

Exclusion Criteria:

* History of clinically significant neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, genitourinary, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
* Known or suspected carcinoma.
* History of hypersensitivity or idiosyncratic reaction to obicetrapib, ezetimibe, or any other drug substances with similar activity.
* History of clinically significant angioedema.
* History of myopathy, rhabdomyolysis, or myalgia, which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
* History of pancreatitis, which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
* History of severe cutaneous adverse reactions (SCARs), Steven-Johnson Syndrome (SJS), toxic epidermal necrolysis (TEN), or drug reaction with eosinophilic and systemic symptoms (DRESS), which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
* Presence of hepatic or renal dysfunction.
* History of malabsorption within the last year or presence of clinically significant gastrointestinal (GI) disease.
* Presence of a medical condition requiring regular medication (prescription and/or over-the-counter) with systemic absorption.
* History of drug or alcohol addiction requiring treatment.
* Positive test result for HIV, Hepatitis B surface antigen, or Hepatitis C antibody.
* Positive test result for urine drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, phencyclidine, and tricyclic antidepressants) or urine cotinine.
* Difficulty fasting or consuming standard meals.
* Use of tobacco or nicotine-containing products within six (6) months prior to the first drug administration.
* Females who:

  * Have used implanted, injected, intravaginal, or intrauterine hormonal contraceptives within six (6) months prior to the first drug administration;
  * Have used oral or transdermal hormonal contraceptives within 21 days prior to the first drug administration;
  * Are pregnant (serum β-hCG consistent with pregnancy); or
  * Are breast-feeding.
* Donation or loss of whole blood (including clinical trials):

  * ≥50 mL and <500 mL within 30 days prior to the first drug administration; or
  * ≥500 mL within 56 days prior to the first drug administration.
* Participation in a clinical trial that involved administration of an investigational medicinal product within 30 days prior to the first drug administration, or recent participation in a clinical investigation that, in the opinion of the Investigator, would jeopardize subject safety or the integrity of the study results.
* On a special diet within 30 days prior to the first drug administration (e.g., liquid, protein, raw food diet).
* Have had a tattoo or body piercing within 30 days prior to the first drug administration.
* Have clinically significant findings in vital signs measurements.
* Have clinically significant findings in a 12-lead ECG.
* Have clinically significant abnormal laboratory values.
* Have significant diseases.
* Use of any of the following within 30 days prior to drug administration:

  * Bile acid sequestrant (e.g., cholestyramine)
  * Cyclosporine
  * Digoxin
  * Drugs that alter GI pH/movement (e.g., omeprazole, ranitidine)
  * Enzyme-modifying drugs known to induce/inhibit hepatic drug metabolism
  * Fibrates (e.g., fenofibrate)
  * Gemfibrozil
  * Glipizide
  * Inducers and inhibitors of breast cancer resistant protein
  * Inducers and inhibitors of CYP3A4
  * Inducers and inhibitors of OATP1B1/OATP1B3
  * Inducers and inhibitors of P-glycoprotein
  * Statin
  * Warfarin
* Have clinically significant findings from a physical examination.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Cmax (Obicetrapib, unconjugated ezetimibe, and ezetimibe glucuronide) | time zero (0) to the time of the last measurable analyte concentration (t), up to 18 days
  Maximum measured analyte concentration
AUCt (Obicetrapib, unconjugated ezetimibe, and ezetimibe glucuronide) | time zero (0) to the time of the last measurable analyte concentration (t)
  The area under the analyte concentration versus time curve
AUCinf (Obicetrapib, unconjugated ezetimibe, and ezetimibe glucuronide) | m time zero to infinity
  The area under the analyte concentration versus time curve

SECONDARY OUTCOMES:
Tmax (Obicetrapib, unconjugated ezetimibe, and ezetimibe glucuronide) | zero (0) to the time of the last measurable analyte concentration (t), up to 18 days
  Time of the maximum measured analyte concentration
Kel (Obicetrapib, unconjugated ezetimibe, and ezetimibe glucuronide) | time zero (0) to the time of the last measurable analyte concentration (t), up to 18 days
  The apparent first-order elimination rate constant
Thalf (Obicetrapib, unconjugated ezetimibe, and ezetimibe glucuronide) | zero (0) to the time of the last measurable analyte concentration (t), up to 18 days
  The apparent elimination half-life
CL/F (Obicetrapib, unconjugated ezetimibe, and ezetimibe glucuronide) | time zero (0) to the time of the last measurable analyte concentration (t), up to 18 days
  Total body clearance
Vd/F (Obicetrapib, unconjugated ezetimibe, and ezetimibe glucuronide) | time zero (0) to the time of the last measurable analyte concentration (t), up to 18 days
  Apparent volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Mark M Feldman, Principal Investigator — Pharma Medica Research, Inc.
Locations (1):
- PharmaMedica Research Inc., Toronto, Ontario, Canada